CLINICAL TRIAL: NCT04221815
Title: IMPact on Revascularization Outcomes of intraVascular Ultrasound Guided Treatment of Complex Lesions and Economic Impact (IMPROVE)
Brief Title: IMPact on Revascularization Outcomes of IVUS Guided Treatment of Complex Lesions and Economic Impact
Acronym: IMPROVE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medstar Health Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IMPROVE
Record Dates: First submitted 2019-12-27; First posted 2020-01-09 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Atherosclerosis
MeSH Terms: conditions — Atherosclerosis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- IVUS guided PCI (Active Comparator): Patients will receive a pre-PCI IVUS, IVUS guided stent sizing and optimization per study protocol, post-PCI IVUS
  Interventions: Device: Eagle Eye Platinum digital IVUS catheter with optional SyncVision; Device: Resolute Onyx Drug Eluting Stent; Device: Onyx Frontier Drug Eluting Stent; Device: Onyx TruStar Drug Eluting Stent; Device: Onyx TruCor Drug Eluting Stent
- Angiographic-guided PCI (Placebo Comparator): Patients will receive angiography guided PCI and angiographic optimization per local standard practice, as well as a post-PCI IVUS blinded to the investigator
  Interventions: Device: Resolute Onyx Drug Eluting Stent; Device: Onyx Frontier Drug Eluting Stent; Device: Onyx TruStar Drug Eluting Stent; Device: Onyx TruCor Drug Eluting Stent

INTERVENTIONS:
Device: Eagle Eye Platinum digital IVUS catheter with optional SyncVision — IVUS catheter
  Arms: IVUS guided PCI
Device: Resolute Onyx Drug Eluting Stent — Stent
Device: Onyx Frontier Drug Eluting Stent — Stent
Device: Onyx TruStar Drug Eluting Stent — Stent
Device: Onyx TruCor Drug Eluting Stent — Stent

SUMMARY:
Intravascular ultrasound (IVUS)-guided percutaneous coronary intervention (PCI) has been shown in clinical trials, registries, and meta-analyses to reduce recurrent events after PCI. This is accomplished by improving the angiographic result with lesion and vessel assessment to guide stent selection and implantation and intravascular imaging following stent implantation to ensure an adequate treatment endpoint has been achieved. Despite extensive literature supporting the use of IVUS in PCI, utilization remains low in the United States. An increasing number of high-risk or complex lesions are being treated with PCI and we hypothesize that the impact of IVUS in these complex lesions will be of increased importance in reducing clinical adverse events while remaining cost effective.

DETAILED DESCRIPTION:
This is a prospective, single-blind clinical investigation randomizing subjects to IVUS-guided coronary stent implantation vs. angiography-guided coronary stent implantation in a 1:1 ratio.

The clinical investigation will be conducted at approximately 120 centers in the US, Canada, and Europe. Approximately 2,500-3,100 randomized subjects and up to 3 roll-in subjects per site will be enrolled in this study. Subjects participating in this clinical investigation will be followed for 2 years. The expected duration of enrollment is approximately 2.5 years. The total duration of the clinical investigation is expected to be approximately 4.5 years.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years at screening
* PCI with stent implantation involving a high risk or complex lesion defined as involving at least one of the following characteristics:
* Chronic total occlusion
* In-stent restenosis
* Severe coronary artery calcification
* Long lesion (≥ 28 mm in length)
* Bifurcation lesion (Any Medina class that involves main branch disease with a side branch ≥2.0 mm)
* Stable angina, unstable angina, or non-ST Elevation myocardial infarction (NSTEMI), undergoing PCI of a single or multivessel coronary artery stenosis
* PCI performed with either angiography alone, or IVUS guidance used

Exclusion Criteria:

* Subjects with acute ST elevation myocardial infarction (STEMI), or cardiogenic shock
* Use of fibrinolytic therapy within 24 hours of PCI
* Planned revascularization of a target vessel as a staged procedure
* Stent thrombosis
* Use of optical coherence tomography (OCT) during the index procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3100 (Estimated)
Dates: Start 2020-10-14 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
IVUS core lab measures final PCI Minimum Stent Area | Intra-procedural
  The imaging primary endpoint is the final post-PCI minimum stent area (MSA) assessed by IVUS in each randomized arm, measured at an independent IVUS core laboratory blinded to treatment assignment. The MSA is an appropriate co-primary imaging endpoint as it is the most consistent and strongest parameter to predict clinical outcomes.11-14 In the present study, after 2,000 subjects are enrolled with the procedure completed, the primary endpoint of MSA will be tested to compare the IVUS-guided and angiography-guided arms. If significantly larger MSA in the IVUS-guided arm is demonstrated, the trial will continue enrolling subjects.
Target vessel failure (TVF) outcomes at 12 months defined as the composite of cardiac death, target vessel related-myocardial infarction (MI), and ischemia-driven target vessel revascularization. | 12 months
  The clinical primary endpoint is target vessel failure (TVF) outcomes at 12 months defined as the composite of cardiac death, target vessel related- myocardial infarction (MI), and target vessel revascularization.

CONTACTS AND LOCATIONS:
Overall Officials: Ron Waksman, MD, Principal Investigator — MedStar Health
Locations (61):
- United States (40):
  - Northwest Medical Center, Tucson, Arizona
  - Central Arkansas Veterans Healthcare System, Little Rock, Arkansas
  - University of California San Deigo, La Jolla, California
  - San Francisco VA Health Care System, San Francisco, California
  - San Antonio Regional Hospital, Upland, California
  - Medstar Washington Hospital Center, Washington D.C., District of Columbia
  - Manatee Memorial Hospital, Bradenton, Florida
  - AdventHealth Orlando, Orlando, Florida
  - Ascension Sacred Heart, Pensacola, Florida
  - AdventHealth Sebring, Sebring, Florida
  - Tampa Cardiovascular/St. Joseph's Hospital, Tampa, Florida
  - Emory, Atlanta, Georgia
  - Atlanta VA Medical Center, Decatur, Georgia
  - Northeast Georgia Medical Center, Gainesville, Georgia
  - Rush University Medial Center, Chicago, Illinois
  - Riverside Medical Center, Kankakee, Illinois
  - Carle Foundation Hospital, Urbana, Illinois
  - MercyOne Iowa Heart Center, Des Moines, Iowa
  - MedStar Union Memorial Hospital, Baltimore, Maryland
  - MedStar Southern Maryland Hospital Center, Clinton, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Baystate Medical Center, Springfield, Massachusetts
  - Ascension St. John, Dearborn, Michigan
  - St. Luke's Hospital of Duluth, Duluth, Minnesota
  - University of Minnesota, Minneapolis, Minnesota
  - Virtua Our Lady of Lourdes Hospital, Camden, New Jersey
  - AtlantiCare Regional Medical Center, Pomona, New Jersey
  - Northwell Health - South Shore University Hospital, Bay Shore, New York
  - NYU Langone Hospital, Brooklyn, New York
  - Northwell Health - North Shore University Hospital, Manhasset, New York
  - Northwell Health - Lennox Hill Hospital, New York, New York
  - St. Francis, Roslyn, New York
  - Good Samaritan University Hospital, West Islip, New York
  - University of North Carolina Rex Hospital, Raleigh, North Carolina
  - The Ohio State University Medical Center, Columbus, Ohio
  - Lehigh Valley Hospital, Allentown, Pennsylvania
  - Seton Medical Center Austin, Austin, Texas
  - Texas Tech University Health Sciences Center, El Paso, Texas
  - Carilion Clinic, Roanoke, Virginia
- Nicosia General Hospital, Nicosia, Cyprus
- Germany (7):
  - Herz-und Diabeteszentrum NRW, Bad Oeynhausen, North Rhine-Westphalia
  - St. Vinzenz Hospital, Cologne, North Rhine-Westphalia
  - Segerberger Kliniken, Bad Segeberg
  - Helios Amper-Klinikum Dachau, Dachau
  - University Medical Center Hamburg-Eppendorf, Hamburg
  - Rheinland Klinikum, Neuss
  - University Medicine Rostock, Rostock
- Greece (3):
  - General Hospital of Athens Hippokration, Athens
  - The University General Hospital of Ioannina, Ioannina
  - Thriassion General Hospital, Magoula
- Israel (2):
  - Shamir Medical Center, Be’er Ya‘aqov
  - Meir Medical Center, Kfar Saba
- Italy (2):
  - University Hospital Careggi, Florence
  - University of Messina, Messina
- Sweden (3):
  - Sahlgrenska University Hospital, Gothenburg
  - Skane University Hospital, Lund
  - Danderyd University Hospital, Stockholm
- United Kingdom (3):
  - Freeman Hospital, Newcastle upon Tyne, Tyne and Wear
  - Leeds General Infirmary, Leeds, West Yorkshire
  - Imperial College Healthcare, London

REFERENCES:
- [Derived] Shlofmitz E, Torguson R, Mintz GS, Zhang C, Sharp A, Hodgson JM, Shah B, Kumar G, Singh J, Inderbitzen B, Weintraub WS, Garcia-Garcia HM, Di Mario C, Waksman R. The IMPact on Revascularization Outcomes of intraVascular ultrasound-guided treatment of complex lesions and Economic impact (IMPROVE) trial: Study design and rationale. Am Heart J. 2020 Oct;228:65-71. doi: 10.1016/j.ahj.2020.08.002. Epub 2020 Aug 8. PMID 32866927